CLINICAL TRIAL: NCT05836974
Title: Performance Evaluation of the ex Utero Cord Blood Collection Technique: Procedure, Quality and Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Nimet Caner, Principal Investigator, Fundacion Dexeus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FSD-BST-2022-08
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Umbilical Cord Blood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ex-utero cord blood collection (Experimental): Ex-utero cord blood collection
  Interventions: Procedure: Ex-utero cord blood collection
- In-utero cord blood collection (Active Comparator): In-utero cord blood collection
  Interventions: Procedure: In-utero cord blood collection

INTERVENTIONS:
Procedure: Ex-utero cord blood collection — SCU units are collected after placental delivery (ex-utero) by trained obstetric personnel. The cord is clamped at one minute postpartum. Once the placenta is expelled, it is rapidly transported to the collection area, which contains supplies and a surgical table designed for ex-utero SCU collection. This table has a top tray supported by an armrest. The placenta is placed on this specially designed tray with a central hole that allows the umbilical cord to hang. Proper asepsis of the cord is first performed with povidone-iodine and then with 70% alcohol. Subsequently, the umbilical vein is cannulated at the most distal point of the placenta, and placental blood is collected by gravity into a sterile bag. Gentle massage can be applied to the placenta to continue draining blood by gravity. If visible blood remains, a second puncture can be made by bringing the needle insertion point closer to the placenta.
  Arms: Ex-utero cord blood collection
Procedure: In-utero cord blood collection — The cord blood is clamped in a delayed modality, defined as after at least 1 minute after delivery. The cord is sterilized, and cord blood is collected using aseptic technique (proper asepsis of the cord is first performed with povidone-iodine and then with 70% alcohol). Blood is allowed to flow by gravity and the needle is removed when blood flow ceases.
  Arms: In-utero cord blood collection

SUMMARY:
Umbilical cord blood (UCB) is used for leukemia patients and other serious blood disorders worldwide. (3) It has also been recently used for other therapeutic applications such as wound treatment, red blood cell transfusion, or cellular or regenerative therapy. Until now, cord blood banks have worked to have many units in reserve to offer maximum compatibility with patients.

The priority is to increase the quality of cord blood by collecting units that have more stem cells with less contamination so that more patients can benefit, that is, improving the efficiency of the process.

The conventional in utero technique allowed for a more rapid diffusion of cord blood donation programs as it does not require accessories or additional personnel to carry it out. The UCB donation program was initiated in Catalonia in 1995, and since then, this has been the technique used (www.bancsang.net/info-corporativa/qui-som). Some comparisons have been made in the scientific literature with the results found . Currently, there are some new applications of UCB that require its use in fresh form, and it would be beneficial to minimize the risk of bacterial contamination that seems to be reduced with ex utero collection. Therefore, the proposition for this study is to confirm equivalence in quality characteristics and create opportunities for its extensive application.

Currently, cord blood donation is offered to all expectant mothers, provided that the donor does not have any medical exclusion. A very small number of the collected units are suitable for clinical use once processed, making donation programs truly inefficient. This inefficiency generates a workload and waste of public resources that are limited and can also cause ethical dilemmas. Therefore, new strategies are needed to increase the efficiency of donation programs. The Blood and Tissue Bank (BST) has an efficiency improvement study underway using the ex-utero collection technique. The development of this methodology will allow later to propose expanded collection methods, such as the simultaneous collection of cord blood and placenta.

The update of new protocols in childbirth care encourages to explore new systematic umbilical cord blood collection methods with the following objectives: to intervene less in the delivery room obtaining products of equal quality and less contamination and to facilitate the simultaneous donation of UCB and placenta in the future. To ensure that the units have maximum quality, both cellular and free of bacteriology, and can be used safely, the investigators propose the implementation of ex utero cord blood collection. The ex-utero UCB collection involves minimal manipulation, allowing for better cord asepsis. After the birth of the baby and cord clamping at one minute, the investigators wait for the delivery of the placenta and proceed to obtain the ex-utero UCB sample. Thanks to this technique, residual cord blood can be obtained, and the placenta can be collected simultaneously, maintaining the same volume as in in utero collection and reducing contamination and hemolysis of the samples.

This technique poses no risk to either the mother or the baby. The ex-utero cord blood collection technique is a validated technique used in different studies.

To verify these data in our environment and propose a change in the cord blood collection strategy in public banks, this study has been designed.

If the investigators demonstrate that this methodology meets quality objectives, similar to the in-utero technique but significantly reducing associated contamination from the delivery field and the presence of hemolysis, the cord blood bank can implement this new systematic method in centers with highly trained collection personnel, releasing obstetric professionals from their intervention in the delivery room and favoring better quality of the products obtained.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Geographical origin and history of known travels
* Absence of potentially transmissible diseases (infectious, hematological, and autoimmune)
* Absence of diseases that can alter prenatal obstetric variables: multiple pregnancy, pregestational diabetes mellitus, intrauterine growth restriction, hypertensive states of pregnancy or chronic arterial hypertension, and fetal pathology.
* Any type of delivery: vaginal delivery and cesarean section.
* Deliveries from week 37 or higher.
* Standardization of the timing of clamping in all cases to one minute.

Exclusion Criteria:

* Pregnant women who meet the exclusion criteria to be cord blood donors.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Weight of cord blood collection | At delivery
  have a minimum weight of 85 grams. Subsequently, the efficiency for certain uses will be evaluated:
  * Biobank for culture media: from 85 to 100 grams
  * Multicomponent cord blood: > 100 grams and less than 1.5 billion leukocytes
  * Transplant: > 100 grams and greater than 15 billion leukocytes

SECONDARY OUTCOMES:
Leukocytes | At delivery
  (White Blood Cells) : cells/µL
Red blood cells | At delivery
  million/µL
Hematocrit | At delivery
  percentage
Platelets | At delivery
  unit of measurement: cells/µ
CD34+ cells | At delivery
  CD34+ cells are hematopoietic stem cells, meaning cells that can differentiate into various types of blood cells. The amount of CD34+ cells in cord blood is an indicator of the sample's ability to generate new blood cells.
Bacteriology | At delivery
  presence/absence. Bacteriology is the study of bacteria present in a biological sample. In the case of cord blood, a bacteriological analysis is performed to detect the presence of bacteria that may affect the sample's quality.
Hemolysis | At delivery
  presence/absence. Hemolysis is the rupture of red blood cells and the release of their contents into the blood. The presence of hemolysis in cord blood may indicate poor sample quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Departamento de Ginecología Obstetricia y Reproducción. Hospital Universitari Dexeus, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Querol S, Gomez SG, Pagliuca A, Torrabadella M, Madrigal JA. Quality rather than quantity: the cord blood bank dilemma. Bone Marrow Transplant. 2010 Jun;45(6):970-8. doi: 10.1038/bmt.2010.7. Epub 2010 Mar 1. PMID 20190835
- [Background] Rocha V, Gluckman E; Eurocord and European Blood and Marrow Transplant Group. Clinical use of umbilical cord blood hematopoietic stem cells. Biol Blood Marrow Transplant. 2006 Jan;12(1 Suppl 1):34-41. doi: 10.1016/j.bbmt.2005.09.006. PMID 16399582
- [Background] Gluckman E. Milestones in umbilical cord blood transplantation. Blood Rev. 2011 Nov;25(6):255-9. doi: 10.1016/j.blre.2011.06.003. Epub 2011 Jul 20. PMID 21764191
- [Background] Solves Alcaina P, Perales Marin A, Mirabet Lis V, Brik Spinelli M, Soler Garcia MA, Roig Oltra R. [Donors selection and retrieval of units in an umbilical cord blood bank]. Med Clin (Barc). 2007 Oct 27;129(15):561-5. doi: 10.1157/13111706. Spanish. PMID 17988611
- [Background] Magalon J, Maiers M, Kurtzberg J, Navarrete C, Rubinstein P, Brown C, Schramm C, Larghero J, Katsahian S, Chabannon C, Picard C, Platz A, Schmidt A, Katz G. Banking or Bankrupting: Strategies for Sustaining the Economic Future of Public Cord Blood Banks. PLoS One. 2015 Dec 1;10(12):e0143440. doi: 10.1371/journal.pone.0143440. eCollection 2015. PMID 26624279
- [Background] Kurtzberg J, Cairo MS, Fraser JK, Baxter-Lowe L, Cohen G, Carter SL, Kernan NA. Results of the cord blood transplantation (COBLT) study unrelated donor banking program. Transfusion. 2005 Jun;45(6):842-55. doi: 10.1111/j.1537-2995.2005.04428.x. PMID 15934981
- [Background] Bart T, Boo M, Balabanova S, Fischer Y, Nicoloso G, Foeken L, Oudshoorn M, Passweg J, Tichelli A, Kindler V, Kurtzberg J, Price T, Regan D, Shpall EJ, Schwabe R. Impact of selection of cord blood units from the United States and swiss registries on the cost of banking operations. Transfus Med Hemother. 2013 Feb;40(1):14-20. doi: 10.1159/000345690. Epub 2013 Jan 7. PMID 23637645
- [Background] Committee Opinion No. 684: Delayed Umbilical Cord Clamping After Birth. Obstet Gynecol. 2017 Jan;129(1):1. doi: 10.1097/AOG.0000000000001860. PMID 28002310
- [Background] Lin X, Torrabadella M, Amat L, Gomez S, Azqueta C, Sanchez M, Cuadras D, Martinez Lorenzo MJ, Brull JM, Gaya A, Cemborain A, Perez Garcia C, Arroyo J, Querol S, Gomez Roig MD. Estimated fetal weight percentile as a tool to predict collection of cord blood units with higher cellular content: implications for prenatal selection of cord blood donors. Transfusion. 2018 Jul;58(7):1732-1738. doi: 10.1111/trf.14651. Epub 2018 May 6. PMID 29732577
- [Background] Vanegas D, Trivino L, Galindo C, Franco L, Salguero G, Camacho B, Perdomo-Arciniegas AM. A new strategy for umbilical cord blood collection developed at the first Colombian public cord blood bank increases total nucleated cell content. Transfusion. 2017 Sep;57(9):2225-2233. doi: 10.1111/trf.14190. Epub 2017 Jun 26. PMID 28653354
- [Background] Solves P, Moraga R, Saucedo E, Perales A, Soler MA, Larrea L, Mirabet V, Planelles D, Carbonell-Uberos F, Monleon J, Planells T, Guillen M, Andres A, Franco E. Comparison between two strategies for umbilical cord blood collection. Bone Marrow Transplant. 2003 Feb;31(4):269-73. doi: 10.1038/sj.bmt.1703809. PMID 12621461
- [Background] Solves P, Moraga R, Mirabet V, Larrea L, Soler MA. In utero or ex utero cord blood collection: an unresolved question. Transfusion. 2003 Aug;43(8):1174-6; author reply 1176. doi: 10.1046/j.1537-2995.2003.00459.x. No abstract available. PMID 12869128
- See also: Related Info — http://www.dexeus.com